CLINICAL TRIAL: NCT04051333
Title: The E-health Application To Modify ORal Energy Intake and Measure Outcomes REmotely in ALS Clinical Trial (EAT MORE2)
Acronym: EAT MORE2
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: ALS Association (Other)
Responsible Party: Principal Investigator, Anne-Marie Alexandra Wills, MD, Assistant Professor of Neurology, Massachusetts General Hospital
Other Study IDs: 2019P001649
Record Dates: First submitted 2019-08-06; First posted 2019-08-09 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ALS Nutrition App (MyDataHelps platform) — We have designed a mobile health app to provide nutritional counseling and to measure disease outcomes both through self-reported questionnaires and through passive data collection.

SUMMARY:
This is phase IIa feasibility and tolerability study of a mobile health (mHealth) application designed to study the effects of remote dietary counseling on disease progression and quality of life. The study will consist of two phases: Part I will consist of building and beta-testing the ALS Nutrition app and Part II will consist of enrolling a larger cohort of users into the app.

DETAILED DESCRIPTION:
The investigators' prior work has shown that nutrition is an important modifiable prognostic factor for ALS disease progression and survival. In the recently completed E-Health Application To Measure Outcomes Remotely (EAT MORE) clinical trial (sponsored by the ALS Association), the investigators found that nutritional counseling supported by a mobile health (mHealth) app was associated with 0.5 points/month slower ALSFRS-R progression (p=0.17) and improved quality of life (p=0.09).

The investigators are now designing an ALS-specific app that can be used by everyone with ALS, including those who do not live near ALS Centers. The app would help to address gaps in the delivery of ALS care by providing nutritional counseling, helping patients to manage and track their disease symptoms, and communicating with their providers. After the initial design has been tested by a group of NEALS patients and their caregivers, the study will advertise the app widely to recruit a larger group of ALS patients to measure nutrition and outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with a diagnosis of ALS (self-reported)
2. Male or female subjects aged 18 years or older.
3. Participants must be capable of providing informed consent and complying with trial procedures.
4. Participants must have access to an iOS or Android device to allow the to download the apps.

Exclusion criteria:

1. Use of a feeding tube (G-tube or J-tube)
2. BMI>30 kg/m2 regardless of weight loss history
3. A history of cardiovascular disease (stroke, myocardial infarction, peripheral vascular disease)
4. A history of diabetes (self-reported)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with ALS without dysphagia, diabetes or cardiovascular disease
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcome Measurement Information System Short Form v1.0 | Change over time over 6 months
  Patient Reported Global Health Questionnaire where the higher the T score the better

SECONDARY OUTCOMES:
ALS Functional Rating Scale-Revised | Change over time over 6 months
  The ALSFRS-R total score ranges from 0-40 with higher scores better

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wills AM, Garry J, Hubbard J, Mezoian T, Breen CT, Ortiz-Miller C, Nalipinski P, Sullivan S, Berry JD, Cudkowicz M, Paganoni S, Chan J, Macklin EA. Nutritional counseling with or without mobile health technology: a randomized open-label standard-of-care-controlled trial in ALS. BMC Neurol. 2019 May 29;19(1):104. doi: 10.1186/s12883-019-1330-6. PMID 31142272